CLINICAL TRIAL: NCT03462212
Title: A Randomized, Molecular Driven Phase II Trial of Carboplatin-Paclitaxel-Bevacizumab vs Carboplatin-Paclitaxel-Bevacizumab-Rucaparib vs Carboplatin-Paclitaxel-Rucaparib, Selected According to HRD Status, in Patients With Advanced (Stage III B-C-IV) Ovarian, Primary Peritoneal and Fallopian Tube Cancer Preceded by a Phase I Dose Escalation Study on Rucaparib-Bevacizumab Combination
Brief Title: Carboplatin-Paclitaxel-Bevacizumab vs Carbo-Pacli-Beva-Rucaparib vs Carbo-Pacli-Ruca, Selected According to HRD Status, in Patients With Advanced Ovarian, Primary Peritoneal and Fallopian Tube Cancer, Preceded by a Phase I Dose Escalation Study on Ruca-Beva Combination
Acronym: MITO25
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other); Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3329
Record Dates: First submitted 2018-02-14; First posted 2018-03-12 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Advanced (Stage IIIB-C-IV) Ovarian, Primary Peritoneal and Fallopian Tube Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Carboplatin; Paclitaxel; Bevacizumab; rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment (Other): Carboplatin AUC 5 + Paclitaxel 175 mg/mq d 1 q 21 for 6 cycles + Bevacizumab 15 mg/kg d 1 q 21 days for 22 cycles (in combination and maintenance)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab
- Carboplatin + Paclitaxel + Bevacizumab + Rucaparib (Experimental): Carboplatin AUC 5 + Paclitaxel 175 mg/mq d1 q 21 days for 6 cycles + Bevacizumab 15 mg/kg d1 q 21 for 22 cycles (in combination and maintenance) + Rucaparib at the dose defined by the Phase I study continuously for 2 years (Rucaparib only in maintenance)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab; Drug: Rucaparib
- Carboplatin + Paclitaxel + Rucaparib (Experimental): Carboplatin AUC 5 + Paclitaxel 175 mg/mq d1 q 21 days for 6 cycles + Rucaparib 600 mg BID continuously for 2 years (Rucaparib only as maintenance).
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Rucaparib

INTERVENTIONS:
Drug: Carboplatin — chemotherapy medication
Drug: Paclitaxel — chemotherapy medication
Drug: Bevacizumab — Angiogenesis inhibitor
  Arms: Carboplatin + Paclitaxel + Bevacizumab + Rucaparib; Standard treatment
Drug: Rucaparib — PARP inhibitor
  Arms: Carboplatin + Paclitaxel + Bevacizumab + Rucaparib; Carboplatin + Paclitaxel + Rucaparib

SUMMARY:
This trial is a randomized, open-label Phase I-2 multi-center study designed to evaluate the effect of Carboplatin-Paclitaxel-Bevacizumab (in combination and maintenance) vs Carboplatin-Paclitaxel-Bevacizumab-Rucaparib (Rucaparib only in maintenance) vs Carboplatin-Paclitaxel-Rucaparib (Rucaparib only in maintenance) on progression-free survival in patients with advanced high grade ovarian cancer treated according to HRD status . The trial will test the hypothesis that Carboplatin-Paclitaxel-Bevacizumab-Rucaparib and the Carboplatin-Paclitaxel-Rucaparib arms will improve the progression-free survival in comparison to standard Carboplatin-Paclitaxel-Bevacizumab in HRD negative (HR proficient) patients and that Carboplatin-Paclitaxel-Bevacizumab-Rucaparib will improve PFS with respect to Carboplatin-Paclitaxel-Rucaparib in HRD positive patients. The randomized phase of the study will be preceded by a single arm Phase I study which will be conducted only in the National Cancer Institute of Milan, aiming at evaluating the MTD of the combination Rucaparib-Bevacizumab. Once the MTD has been reached, the randomized study will start.

DETAILED DESCRIPTION:
Phase I study design:

This is a single-centre, Phase I, open-label, dose-escalation study to evaluate the safety and tolerability of bevacizumab-rucaparib combination and determine the MTD in patients with advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer.

The dose of bevacizumab is fixed in cohort 1, 2 and 3 of the study at 15mg/kg, q 3 weekly.

The dose of rucaparib is evaluated in three cohorts (400 mg BID; 500 mg BID; 600 mg BID).

This trial will enroll at least 3 patients in cohort 1 with dose escalation to rucaparib 500 mg from cohort 1 to 2. Cohort 2 will enroll at least 3 patients with dose escalation to rucaparib 600 mg from cohort 2 to 3.

The standard 3+3 design will be used. Patients will be enrolled in cohort of 3 patients, if no DLT event will be reported among the first 3 patients, a second cohort will be enrolled at the upper dose level. If 1 DLT event is registered in the first cohort, other 3 patients will be enrolled at the same dose.

Phase II study design:

Eligible patients with histological documented high grade Stage IIIB-IIIC-IV ovarian cancer (regardless of residual tumor) will be randomized 1:1:1 according to a molecular driven treatment.

HRD positive patients:

* ARM B: Carboplatin AUC 5 + Paclitaxel 175 mg/m2 q 21 for 6 cycles followed by Rucaparib 600 mg BID q 28 for 24 cycles as maintenance
* ARM C: Carboplatin AUC 5+ Paclitaxel 175 mg/m2 q 21 + Bevacizumab 15 mg/kg for 6 cycles followed by Bevacizumab 15 mg/kg q 21 days for 16 cycles (Bevacizumab will start from Cycle 2) + Rucaparib 500 mg part BID q 28 for 24 cycles as maintenance

HRD negative patients:

* ARM A: Carboplatin AUC 5 + Paclitaxel 175 mg/m2 q 21 + Bevacizumab 15 mg/kg for 6 cycles followed by Bevacizumab 15 mg/kg q 21 for 16 cycles (Bevacizumab will start from Cycle 2)
* ARM B: Carboplatin AUC 5 + Paclitaxel 175 mg/m2 q 21 for 6 cycles followed by Rucaparib 600 mg BID q 28 for 24 cycles as maintenance

Stratification factors are:

* Residual tumor at primary surgery (RT=0 vs RT> 0)
* Neoadiuvant chemotherapy (Yes or not)

ELIGIBILITY:
Inclusion Criteria:

1. Women aged >=18 years at the time of study inclusion;
2. Patients with newly diagnosed, histologically confirmed, high grade serous, high grade endometrioid, FIGO stage IIIB-C-IV epithelial ovarian cancer, primary peritoneal cancer and / or Fallopian-tube cancer. Patients with mixed histology (carcinosarcoma) are eligible providing that high grade tumor represent more than 50% of the total histology.

   Stage III patients should have had one attempt at optimal debulking surgery (upfront or interval debulking). Stage IV patients must have had either a biopsy and/or upfront or interval debulking surgery;
3. Archival tumor tissue available. At progression fresh biopsy is optional for patients willing to submit ;
4. ECOG Performance Status of 0-1;
5. Measurable and not measurable disease;
6. Adequate renal and hepatic function, defined as:

   * Total serum bilirubin ≤ 1.5 institutional ULN unless patient has Gilbert's syndrome in which case total serum bilirubin must be <2 ULN for the institution AST and/or ALT ≤ 2.5 x ULN for the institution. (or ≤ 5 x ULN if liver metastases are present);
   * Alkaline phosphatase < 1.5 x ULN for the institution (if > 1.5 x ULN, then alkaline phosphatase liver fraction must be < 1.5 ULN)
   * Serum creatinine ≤ 1.5 x ULN for the institution (or calculated creatinine clearance ≥ 45 mL/min/1.73 m2);
7. Adequate bone marrow function, defined as:

   * Total leukocytes 2.5 x 109/L;
   * ANC 1.5 x 109/L;
   * Platelet count 100 x 109/L;
8. Able to understand and give written informed consent;
9. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

1. Women who are pregnant or lactating;
2. Presence of brain or other central nervous system metastases, not adequately controlled by treatment;
3. Prior Anticancer treatment;
4. Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 3 weeks prior to randomization;
5. Another primary malignancy except for:

   1. Curatively treated non-melanoma skin cancer;
   2. Breast cancer treated curatively ≥5 years ago, or other solid tumor treated curatively ≥5 years ago, without evidence of recurrence;
   3. Synchronous endometrioid endometrial cancer (except for Stage 1A G1/G2);
6. Known active HIV, hepatitis B or C infection;
7. Concurrent treatment with immunosuppressive or investigational agents;
8. History or evidence of thrombotic or hemorrhagic disorders; including cerebrovascular accident (CVA) / stroke or transient ischemic attack (TIA) or subarachnoid haemorrhage within _6 months prior to the first study treatment);
9. Clinically significant (i.e. active) cardiovascular disease, including:

   * Myocardial infarction or unstable angina within _6 months prior to the first study treatment;
   * New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF);
   * Serious cardiac arrhythmia requiring medication (with the exception of atrial fibrillation or paroxysmal supraventricular tachycardia);
   * Peripheral vascular disease > grade 3 (i.e.symptomatic and interfering with activities of daily living requiring repair or revision);
10. Serious active infection requiring i.v. antibiotics at enrolment;
11. Known hypersensitivity to any of the study drugs or excipients (including cremophor and hamster Ovary cell products);
12. Evidence of any other medical conditions (such as psychiatric illness, peptic ulcer, etc.), physical examination or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment related complications;
13. Prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with absorption of study drug;
14. Received administration of strong CYP1A2 or CYP3A4 inhibitors ≤7 days prior to first dose of Rucaparib or have on-going requirements for these medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 290 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Phase I Primary Objective: MTD | 4 months
  To identify the Maximum Tolerated Dose (MTD) of the combination Rucaparib-Bevacizumab in stage IIIB-C-IV ovarian cancer patients
Phase II Primary Objective: PFS | from the date of randomization to the date of documented progression disease, recurrence or death (whichever occurs first), assessed up to 64 months
  To compare progression-free survival (PFS) of patients with advanced ovarian, primary peritoneal and Fallopian tube cancer when treated with Carboplatin-Paclitaxel-Bevacizumab vs Carboplatin-Paclitaxel-Bevacizumab-Rucaparib vs carboplatin-Paclitaxel-Rucaparib according to Homologous Recombination Deficient (HRD) status.

SECONDARY OUTCOMES:
Phase I Secondary Objectives: toxicity of the Rucaparib-Bevacizumab combination in terms of haematologic and non haematologic events | 4 months
  Toxicity will be evaluated according to U.S. NCI Common Toxicity Criteria version 4.03
Phase I Secondary Objectives: maximum plasma concentration (Cmax at Steady State) of Rucaparib | will be evaluated during cycle 1, on days -7,1,21
  The evaluation of the effect of bevacizumab on rucaparib Cmax at SS will be performed by comparing (in each individual patient) the Cmax during cycle 1, on days 1 and 21, with the Cmax obtained on day -7 in which only Rucaparib will be administered. For these parameters, the following descriptive statistics will be calculated: mean, standard deviation, coefficient of variation, median, and geometric mean.
Phase I Secondary Objectives: minimal plasma concentration (Cmin at Steady State) of Rucaparib | will be evaluated during cycle 1, on days -7,1,21
  The evaluation of the effect of bevacizumab on rucaparib Cmin at SS will be performed by comparing (in each individual patient) the Cmin during cycle 1, on days 1 and 21, with the Cmax obtained on day -7 in which only Rucaparib will be administered. For these parameters, the following descriptive statistics will be calculated: mean, standard deviation, coefficient of variation, median, and geometric mean.
Phase I Secondary Objectives: Area Under Curve (AUC) | will be evaluated during cycle 1, on days -7,1,21
  The evaluation of the effect of bevacizumab on rucaparib AUC will be performed by comparing (in each individual patient) during cycle 1, on days 1 and 21, rucaparib AUC with AUC obtained on day -7 in which only Rucaparib will be administered. For this parameters, the following descriptive statistics will be calculated: mean, standard deviation, coefficient of variation, median, and geometric mean.
Phase I Secondary Objectives: Cmax | will be evaluated during cycle 1, on day1
  The evaluation of the effect of bevacizumab on rucaparib Cmax will be performed by measuring the maximum seric concentration of drug. For this parameter, the following descriptive statistics will be calculated: mean, standard deviation, coefficient of variation, median, and geometric mean.
Phase I Secondary Objectives: Tmax | will be evaluated during cycle 1, on day1
  The evaluation of the effect of bevacizumab on rucaparib will be performed by measuring the amount of time that the drug is present at the maximum concentration in serum. For this parameter, the following descriptive statistics will be calculated: mean, standard deviation, coefficient of variation, median, and geometric mean.
Phase I Secondary Objectives: AUC (0-24h) | will be evaluated during cycle 1, on day1
  The evaluation of the effect of bevacizumab on rucaparib will be performed by measuring the AUC during 24 h. For this parameter, the following descriptive statistics will be calculated: mean, standard deviation, coefficient of variation, median, and geometric mean.
Phase II Secondary Objectives: OS | from the date of randomization to the date of death, assessed up to 64 months
  Overall survival
Phase II Secondary Objectives: PFS2 | from randomisation to second objective disease progression or death, assessed up to 64 months
  Progression-free survival 2
Phase II Secondary Objectives: TFST | from randomisation to the initiation of first subsequent therapy or death of patients, assessed up to 64 months
  Time to first subsequent therapy
Phase II Secondary Objectives: TSST | from randomisation to the initiation of second subsequent therapy or death, assessed up to 64 months
  Time to second subsequent therapy
Phase II Secondary Objectives: ORR | 64 months
  Overall response rate
Phase II Secondary Objectives: Safety and tolerability | 64 months
  Safety and tolerability will be evaluated by U.S. National Cancer Institute Common Toxicity Criteria Adverse Event (NCI CTCAE) version 4.03 and the number of dose reductions
Phase II Secondary Objectives: PRO for PHYSICAL WELL-BEING | 64 months
  Patient-reported outcome (PRO) of disease-related symptoms will be recorded utilizing the disease-related symptoms - physical (DRS-P) subscale of the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCN-FACT) FACT-Ovarian Symptom Index 18 (FOSI-18) changes and using Euro-Quality of Life 5D (EQ-5D) tool (Appendix A).
Phase II Secondary Objectives: PRO for SOCIAL/FAMILY WELL-BEING | 64 months
  Patient-reported outcome (PRO) of disease-related symptoms will be recorded utilizing the disease-related symptoms - physical (DRS-P) subscale of the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCN-FACT) FACT-Ovarian Symptom Index 18 (FOSI-18) changes and using Euro-Quality of Life 5D (EQ-5D) tool (Appendix A).
Phase II Secondary Objectives: PRO for EMOTIONAL WELL-BEING | 64 months
  Patient-reported outcome (PRO) of disease-related symptoms will be recorded utilizing the disease-related symptoms - physical (DRS-P) subscale of the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCN-FACT) FACT-Ovarian Symptom Index 18 (FOSI-18) changes and using Euro-Quality of Life 5D (EQ-5D) tool (Appendix A).
Phase II Secondary Objectives: PRO for FUNCTIONAL WELL-BEING | 64 months
  Patient-reported outcome (PRO) of disease-related symptoms will be recorded utilizing the disease-related symptoms - physical (DRS-P) subscale of the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy (NCCN-FACT) FACT-Ovarian Symptom Index 18 (FOSI-18) changes and using Euro-Quality of Life 5D (EQ-5D) tool (Appendix A).

CONTACTS AND LOCATIONS:
Overall Officials: Domenica Lorusso, Prof., Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (7):
- Italy (7):
  - Ospedale Mater Salutis, Legnago
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Naples
  - Azienda Ospedaliera di Perugia, Perugia
  - Nuovo Ospedale degli Infermi, Ponderano
  - Fondazione Policlinico Universitario A.Gemelli IRCCS, Rome
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia - IRCCS, Turin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Bono JS, Mina LA, Gonzalez M, Curtin NJ, Wang E, Henshaw JW, et al. First-in-human trial of novel oral PARP inhibitor BMN 673 in patients with solid tumors. J Clin Oncol. 2013;31(suppl):2580.
- [Background] Iain A. McNeish, Amit M. Oza, Robert L. Coleman, et al. Results of ARIEL2: A Phase II trial to prospectively identify ovarian cancer patients likely to respond to rucaparib using tumor genetic analysis. J Clin Oncol 33, 2015 (suppl; abstr 5508)
- [Background] Gourley, C. McCavigan, A Perren, T et al Molecular subgroup of high-grade serous ovarian cancer (HGSOC) as a predictor of outcome following bevacizumab. Abstract 5502 ASC0 2014
- [Result] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Result] Chan JK, Cheung MK, Husain A, Teng NN, West D, Whittemore AS, Berek JS, Osann K. Patterns and progress in ovarian cancer over 14 years. Obstet Gynecol. 2006 Sep;108(3 Pt 1):521-8. doi: 10.1097/01.AOG.0000231680.58221.a7. PMID 16946210
- [Result] Engel J, Eckel R, Schubert-Fritschle G, Kerr J, Kuhn W, Diebold J, Kimmig R, Rehbock J, Holzel D. Moderate progress for ovarian cancer in the last 20 years: prolongation of survival, but no improvement in the cure rate. Eur J Cancer. 2002 Dec;38(18):2435-45. doi: 10.1016/s0959-8049(02)00495-1. PMID 12460789
- [Result] Harries M, Gore M. Part I: chemotherapy for epithelial ovarian cancer-treatment at first diagnosis. Lancet Oncol. 2002 Sep;3(9):529-36. doi: 10.1016/s1470-2045(02)00846-x. PMID 12217790
- [Result] International Collaborative Ovarian Neoplasm Group. Paclitaxel plus carboplatin versus standard chemotherapy with either single-agent carboplatin or cyclophosphamide, doxorubicin, and cisplatin in women with ovarian cancer: the ICON3 randomised trial. Lancet. 2002 Aug 17;360(9332):505-15. doi: 10.1016/S0140-6736(02)09738-6. PMID 12241653
- [Result] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Result] McGuire WP, Hoskins WJ, Brady MF, Kucera PR, Partridge EE, Look KY, Clarke-Pearson DL, Davidson M. Cyclophosphamide and cisplatin compared with paclitaxel and cisplatin in patients with stage III and stage IV ovarian cancer. N Engl J Med. 1996 Jan 4;334(1):1-6. doi: 10.1056/NEJM199601043340101. PMID 7494563
- [Result] Muggia FM, Braly PS, Brady MF, Sutton G, Niemann TH, Lentz SL, Alvarez RD, Kucera PR, Small JM. Phase III randomized study of cisplatin versus paclitaxel versus cisplatin and paclitaxel in patients with suboptimal stage III or IV ovarian cancer: a gynecologic oncology group study. J Clin Oncol. 2000 Jan;18(1):106-15. doi: 10.1200/JCO.2000.18.1.106. PMID 10623700
- [Result] Piccart MJ, Bertelsen K, James K, Cassidy J, Mangioni C, Simonsen E, Stuart G, Kaye S, Vergote I, Blom R, Grimshaw R, Atkinson RJ, Swenerton KD, Trope C, Nardi M, Kaern J, Tumolo S, Timmers P, Roy JA, Lhoas F, Lindvall B, Bacon M, Birt A, Andersen JE, Zee B, Paul J, Baron B, Pecorelli S. Randomized intergroup trial of cisplatin-paclitaxel versus cisplatin-cyclophosphamide in women with advanced epithelial ovarian cancer: three-year results. J Natl Cancer Inst. 2000 May 3;92(9):699-708. doi: 10.1093/jnci/92.9.699. PMID 10793106
- [Result] Spannuth WA, Sood AK, Coleman RL. Angiogenesis as a strategic target for ovarian cancer therapy. Nat Clin Pract Oncol. 2008 Apr;5(4):194-204. doi: 10.1038/ncponc1051. Epub 2008 Feb 12. PMID 18268546
- [Result] du Bois A, Quinn M, Thigpen T, Vermorken J, Avall-Lundqvist E, Bookman M, Bowtell D, Brady M, Casado A, Cervantes A, Eisenhauer E, Friedlaender M, Fujiwara K, Grenman S, Guastalla JP, Harper P, Hogberg T, Kaye S, Kitchener H, Kristensen G, Mannel R, Meier W, Miller B, Neijt JP, Oza A, Ozols R, Parmar M, Pecorelli S, Pfisterer J, Poveda A, Provencher D, Pujade-Lauraine E, Randall M, Rochon J, Rustin G, Sagae S, Stehman F, Stuart G, Trimble E, Vasey P, Vergote I, Verheijen R, Wagner U; Gynecologic Cancer Intergroup; AGO-OVAR; ANZGOG; EORTC; GEICO; GINECO; GOG; JGOG; MRC/NCRI; NCIC-CTG; NCI-US; NSGO; RTOG; SGCTG; IGCS; Organizational team of the two prior International OCCC. 2004 consensus statements on the management of ovarian cancer: final document of the 3rd International Gynecologic Cancer Intergroup Ovarian Cancer Consensus Conference (GCIG OCCC 2004). Ann Oncol. 2005;16 Suppl 8:viii7-viii12. doi: 10.1093/annonc/mdi961. No abstract available. PMID 16239238
- [Result] Presta LG, Chen H, O'Connor SJ, Chisholm V, Meng YG, Krummen L, Winkler M, Ferrara N. Humanization of an anti-vascular endothelial growth factor monoclonal antibody for the therapy of solid tumors and other disorders. Cancer Res. 1997 Oct 15;57(20):4593-9. PMID 9377574
- [Result] Jain RK. Normalizing tumor vasculature with anti-angiogenic therapy: a new paradigm for combination therapy. Nat Med. 2001 Sep;7(9):987-9. doi: 10.1038/nm0901-987. No abstract available. PMID 11533692
- [Result] Sweeney CJ, Miller KD, Sissons SE, Nozaki S, Heilman DK, Shen J, Sledge GW Jr. The antiangiogenic property of docetaxel is synergistic with a recombinant humanized monoclonal antibody against vascular endothelial growth factor or 2-methoxyestradiol but antagonized by endothelial growth factors. Cancer Res. 2001 Apr 15;61(8):3369-72. PMID 11309294
- [Result] Borgstrom P, Gold DP, Hillan KJ, Ferrara N. Importance of VEGF for breast cancer angiogenesis in vivo: implications from intravital microscopy of combination treatments with an anti-VEGF neutralizing monoclonal antibody and doxorubicin. Anticancer Res. 1999 Sep-Oct;19(5B):4203-14. PMID 10628376
- [Result] Yuan F, Chen Y, Dellian M, Safabakhsh N, Ferrara N, Jain RK. Time-dependent vascular regression and permeability changes in established human tumor xenografts induced by an anti-vascular endothelial growth factor/vascular permeability factor antibody. Proc Natl Acad Sci U S A. 1996 Dec 10;93(25):14765-70. doi: 10.1073/pnas.93.25.14765. PMID 8962129
- [Result] Kanai T, Konno H, Tanaka T, Baba M, Matsumoto K, Nakamura S, Yukita A, Asano M, Suzuki H, Baba S. Anti-tumor and anti-metastatic effects of human-vascular-endothelial-growth-factor-neutralizing antibody on human colon and gastric carcinoma xenotransplanted orthotopically into nude mice. Int J Cancer. 1998 Sep 11;77(6):933-6. doi: 10.1002/(sici)1097-0215(19980911)77:63.0.co;2-0. PMID 9714067
- [Result] Burger RA, Brady MF, Bookman MA, Fleming GF, Monk BJ, Huang H, Mannel RS, Homesley HD, Fowler J, Greer BE, Boente M, Birrer MJ, Liang SX; Gynecologic Oncology Group. Incorporation of bevacizumab in the primary treatment of ovarian cancer. N Engl J Med. 2011 Dec 29;365(26):2473-83. doi: 10.1056/NEJMoa1104390. PMID 22204724
- [Result] Perren TJ, Swart AM, Pfisterer J, Ledermann JA, Pujade-Lauraine E, Kristensen G, Carey MS, Beale P, Cervantes A, Kurzeder C, du Bois A, Sehouli J, Kimmig R, Stahle A, Collinson F, Essapen S, Gourley C, Lortholary A, Selle F, Mirza MR, Leminen A, Plante M, Stark D, Qian W, Parmar MK, Oza AM; ICON7 Investigators. A phase 3 trial of bevacizumab in ovarian cancer. N Engl J Med. 2011 Dec 29;365(26):2484-96. doi: 10.1056/NEJMoa1103799. PMID 22204725
- [Result] Cannistra SA, Matulonis UA, Penson RT, Hambleton J, Dupont J, Mackey H, Douglas J, Burger RA, Armstrong D, Wenham R, McGuire W. Phase II study of bevacizumab in patients with platinum-resistant ovarian cancer or peritoneal serous cancer. J Clin Oncol. 2007 Nov 20;25(33):5180-6. doi: 10.1200/JCO.2007.12.0782. PMID 18024865
- [Result] Pujade-Lauraine E, Hilpert F, Weber B, Reuss A, Poveda A, Kristensen G, Sorio R, Vergote I, Witteveen P, Bamias A, Pereira D, Wimberger P, Oaknin A, Mirza MR, Follana P, Bollag D, Ray-Coquard I. Bevacizumab combined with chemotherapy for platinum-resistant recurrent ovarian cancer: The AURELIA open-label randomized phase III trial. J Clin Oncol. 2014 May 1;32(13):1302-8. doi: 10.1200/JCO.2013.51.4489. Epub 2014 Mar 17. PMID 24637997
- [Result] Bryant HE, Schultz N, Thomas HD, Parker KM, Flower D, Lopez E, Kyle S, Meuth M, Curtin NJ, Helleday T. Specific killing of BRCA2-deficient tumours with inhibitors of poly(ADP-ribose) polymerase. Nature. 2005 Apr 14;434(7035):913-7. doi: 10.1038/nature03443. PMID 15829966
- [Result] Farmer H, McCabe N, Lord CJ, Tutt AN, Johnson DA, Richardson TB, Santarosa M, Dillon KJ, Hickson I, Knights C, Martin NM, Jackson SP, Smith GC, Ashworth A. Targeting the DNA repair defect in BRCA mutant cells as a therapeutic strategy. Nature. 2005 Apr 14;434(7035):917-21. doi: 10.1038/nature03445. PMID 15829967
- [Result] Alsop K, Fereday S, Meldrum C, deFazio A, Emmanuel C, George J, Dobrovic A, Birrer MJ, Webb PM, Stewart C, Friedlander M, Fox S, Bowtell D, Mitchell G. BRCA mutation frequency and patterns of treatment response in BRCA mutation-positive women with ovarian cancer: a report from the Australian Ovarian Cancer Study Group. J Clin Oncol. 2012 Jul 20;30(21):2654-63. doi: 10.1200/JCO.2011.39.8545. Epub 2012 Jun 18. PMID 22711857
- [Result] Cancer Genome Atlas Research Network. Integrated genomic analyses of ovarian carcinoma. Nature. 2011 Jun 29;474(7353):609-15. doi: 10.1038/nature10166. PMID 21720365
- [Result] Hennessy BT, Timms KM, Carey MS, Gutin A, Meyer LA, Flake DD 2nd, Abkevich V, Potter J, Pruss D, Glenn P, Li Y, Li J, Gonzalez-Angulo AM, McCune KS, Markman M, Broaddus RR, Lanchbury JS, Lu KH, Mills GB. Somatic mutations in BRCA1 and BRCA2 could expand the number of patients that benefit from poly (ADP ribose) polymerase inhibitors in ovarian cancer. J Clin Oncol. 2010 Aug 1;28(22):3570-6. doi: 10.1200/JCO.2009.27.2997. Epub 2010 Jul 6. PMID 20606085
- [Result] Shinohara A, Ogawa H, Ogawa T. Rad51 protein involved in repair and recombination in S. cerevisiae is a RecA-like protein. Cell. 1992 May 1;69(3):457-70. doi: 10.1016/0092-8674(92)90447-k. PMID 1581961
- [Result] Kurumizaka H, Ikawa S, Nakada M, Eda K, Kagawa W, Takata M, Takeda S, Yokoyama S, Shibata T. Homologous-pairing activity of the human DNA-repair proteins Xrcc3.Rad51C. Proc Natl Acad Sci U S A. 2001 May 8;98(10):5538-43. doi: 10.1073/pnas.091603098. Epub 2001 May 1. PMID 11331762
- [Result] Lisby M, Rothstein R, Mortensen UH. Rad52 forms DNA repair and recombination centers during S phase. Proc Natl Acad Sci U S A. 2001 Jul 17;98(15):8276-82. doi: 10.1073/pnas.121006298. PMID 11459964
- [Result] Sigurdsson S, Van Komen S, Petukhova G, Sung P. Homologous DNA pairing by human recombination factors Rad51 and Rad54. J Biol Chem. 2002 Nov 8;277(45):42790-4. doi: 10.1074/jbc.M208004200. Epub 2002 Aug 29. PMID 12205100
- [Result] Yang YG, Herceg Z, Nakanishi K, Demuth I, Piccoli C, Michelon J, Hildebrand G, Jasin M, Digweed M, Wang ZQ. The Fanconi anemia group A protein modulates homologous repair of DNA double-strand breaks in mammalian cells. Carcinogenesis. 2005 Oct;26(10):1731-40. doi: 10.1093/carcin/bgi134. Epub 2005 May 19. PMID 15905196
- [Result] Niedzwiedz W, Mosedale G, Johnson M, Ong CY, Pace P, Patel KJ. The Fanconi anaemia gene FANCC promotes homologous recombination and error-prone DNA repair. Mol Cell. 2004 Aug 27;15(4):607-20. doi: 10.1016/j.molcel.2004.08.009. PMID 15327776
- [Result] Beucher A, Birraux J, Tchouandong L, Barton O, Shibata A, Conrad S, Goodarzi AA, Krempler A, Jeggo PA, Lobrich M. ATM and Artemis promote homologous recombination of radiation-induced DNA double-strand breaks in G2. EMBO J. 2009 Nov 4;28(21):3413-27. doi: 10.1038/emboj.2009.276. Epub 2009 Sep 24. PMID 19779458
- [Result] Chanoux RA, Yin B, Urtishak KA, Asare A, Bassing CH, Brown EJ. ATR and H2AX cooperate in maintaining genome stability under replication stress. J Biol Chem. 2009 Feb 27;284(9):5994-6003. doi: 10.1074/jbc.M806739200. Epub 2008 Dec 2. PMID 19049966
- [Result] Sorensen CS, Hansen LT, Dziegielewski J, Syljuasen RG, Lundin C, Bartek J, Helleday T. The cell-cycle checkpoint kinase Chk1 is required for mammalian homologous recombination repair. Nat Cell Biol. 2005 Feb;7(2):195-201. doi: 10.1038/ncb1212. Epub 2005 Jan 23. PMID 15665856
- [Result] Zhang J, Willers H, Feng Z, Ghosh JC, Kim S, Weaver DT, Chung JH, Powell SN, Xia F. Chk2 phosphorylation of BRCA1 regulates DNA double-strand break repair. Mol Cell Biol. 2004 Jan;24(2):708-18. doi: 10.1128/MCB.24.2.708-718.2004. PMID 14701743
- [Result] Abkevich V, Timms KM, Hennessy BT, Potter J, Carey MS, Meyer LA, Smith-McCune K, Broaddus R, Lu KH, Chen J, Tran TV, Williams D, Iliev D, Jammulapati S, FitzGerald LM, Krivak T, DeLoia JA, Gutin A, Mills GB, Lanchbury JS. Patterns of genomic loss of heterozygosity predict homologous recombination repair defects in epithelial ovarian cancer. Br J Cancer. 2012 Nov 6;107(10):1776-82. doi: 10.1038/bjc.2012.451. Epub 2012 Oct 9. PMID 23047548
- [Result] Wang ZC, Birkbak NJ, Culhane AC, Drapkin R, Fatima A, Tian R, Schwede M, Alsop K, Daniels KE, Piao H, Liu J, Etemadmoghadam D, Miron A, Salvesen HB, Mitchell G, DeFazio A, Quackenbush J, Berkowitz RS, Iglehart JD, Bowtell DD; Australian Ovarian Cancer Study Group; Matulonis UA. Profiles of genomic instability in high-grade serous ovarian cancer predict treatment outcome. Clin Cancer Res. 2012 Oct 15;18(20):5806-15. doi: 10.1158/1078-0432.CCR-12-0857. Epub 2012 Aug 21. PMID 22912389
- [Result] Audeh MW, Carmichael J, Penson RT, Friedlander M, Powell B, Bell-McGuinn KM, Scott C, Weitzel JN, Oaknin A, Loman N, Lu K, Schmutzler RK, Matulonis U, Wickens M, Tutt A. Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with BRCA1 or BRCA2 mutations and recurrent ovarian cancer: a proof-of-concept trial. Lancet. 2010 Jul 24;376(9737):245-51. doi: 10.1016/S0140-6736(10)60893-8. Epub 2010 Jul 6. PMID 20609468
- [Result] Tutt A, Robson M, Garber JE, Domchek SM, Audeh MW, Weitzel JN, Friedlander M, Arun B, Loman N, Schmutzler RK, Wardley A, Mitchell G, Earl H, Wickens M, Carmichael J. Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with BRCA1 or BRCA2 mutations and advanced breast cancer: a proof-of-concept trial. Lancet. 2010 Jul 24;376(9737):235-44. doi: 10.1016/S0140-6736(10)60892-6. Epub 2010 Jul 6. PMID 20609467
- [Result] Gelmon KA, Tischkowitz M, Mackay H, Swenerton K, Robidoux A, Tonkin K, Hirte H, Huntsman D, Clemons M, Gilks B, Yerushalmi R, Macpherson E, Carmichael J, Oza A. Olaparib in patients with recurrent high-grade serous or poorly differentiated ovarian carcinoma or triple-negative breast cancer: a phase 2, multicentre, open-label, non-randomised study. Lancet Oncol. 2011 Sep;12(9):852-61. doi: 10.1016/S1470-2045(11)70214-5. Epub 2011 Aug 19. PMID 21862407
- [Result] Kaye SB, Lubinski J, Matulonis U, Ang JE, Gourley C, Karlan BY, Amnon A, Bell-McGuinn KM, Chen LM, Friedlander M, Safra T, Vergote I, Wickens M, Lowe ES, Carmichael J, Kaufman B. Phase II, open-label, randomized, multicenter study comparing the efficacy and safety of olaparib, a poly (ADP-ribose) polymerase inhibitor, and pegylated liposomal doxorubicin in patients with BRCA1 or BRCA2 mutations and recurrent ovarian cancer. J Clin Oncol. 2012 Feb 1;30(4):372-9. doi: 10.1200/JCO.2011.36.9215. Epub 2011 Dec 27. PMID 22203755
- [Result] Ledermann J, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott C, Meier W, Shapira-Frommer R, Safra T, Matei D, Macpherson E, Watkins C, Carmichael J, Matulonis U. Olaparib maintenance therapy in platinum-sensitive relapsed ovarian cancer. N Engl J Med. 2012 Apr 12;366(15):1382-92. doi: 10.1056/NEJMoa1105535. Epub 2012 Mar 27. PMID 22452356
- [Result] Ledermann J, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott CL, Meier W, Shapira-Frommer R, Safra T, Matei D, Fielding A, Spencer S, Dougherty B, Orr M, Hodgson D, Barrett JC, Matulonis U. Olaparib maintenance therapy in patients with platinum-sensitive relapsed serous ovarian cancer: a preplanned retrospective analysis of outcomes by BRCA status in a randomised phase 2 trial. Lancet Oncol. 2014 Jul;15(8):852-61. doi: 10.1016/S1470-2045(14)70228-1. Epub 2014 May 31. PMID 24882434
- [Result] Sandhu SK, Schelman WR, Wilding G, Moreno V, Baird RD, Miranda S, Hylands L, Riisnaes R, Forster M, Omlin A, Kreischer N, Thway K, Gevensleben H, Sun L, Loughney J, Chatterjee M, Toniatti C, Carpenter CL, Iannone R, Kaye SB, de Bono JS, Wenham RM. The poly(ADP-ribose) polymerase inhibitor niraparib (MK4827) in BRCA mutation carriers and patients with sporadic cancer: a phase 1 dose-escalation trial. Lancet Oncol. 2013 Aug;14(9):882-92. doi: 10.1016/S1470-2045(13)70240-7. Epub 2013 Jun 28. PMID 23810788
- [Result] McCabe N, Turner NC, Lord CJ, Kluzek K, Bialkowska A, Swift S, Giavara S, O'Connor MJ, Tutt AN, Zdzienicka MZ, Smith GC, Ashworth A. Deficiency in the repair of DNA damage by homologous recombination and sensitivity to poly(ADP-ribose) polymerase inhibition. Cancer Res. 2006 Aug 15;66(16):8109-15. doi: 10.1158/0008-5472.CAN-06-0140. PMID 16912188
- [Result] Murai J, Huang SY, Das BB, Renaud A, Zhang Y, Doroshow JH, Ji J, Takeda S, Pommier Y. Trapping of PARP1 and PARP2 by Clinical PARP Inhibitors. Cancer Res. 2012 Nov 1;72(21):5588-99. doi: 10.1158/0008-5472.CAN-12-2753. PMID 23118055
- [Result] Min A, Im SA, Yoon YK, Song SH, Nam HJ, Hur HS, Kim HP, Lee KH, Han SW, Oh DY, Kim TY, O'Connor MJ, Kim WH, Bang YJ. RAD51C-deficient cancer cells are highly sensitive to the PARP inhibitor olaparib. Mol Cancer Ther. 2013 Jun;12(6):865-77. doi: 10.1158/1535-7163.MCT-12-0950. Epub 2013 Mar 19. PMID 23512992
- [Result] Gottipati P, Vischioni B, Schultz N, Solomons J, Bryant HE, Djureinovic T, Issaeva N, Sleeth K, Sharma RA, Helleday T. Poly(ADP-ribose) polymerase is hyperactivated in homologous recombination-defective cells. Cancer Res. 2010 Jul 1;70(13):5389-98. doi: 10.1158/0008-5472.CAN-09-4716. Epub 2010 Jun 15. PMID 20551068
- [Result] Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, Mortimer P, Swaisland H, Lau A, O'Connor MJ, Ashworth A, Carmichael J, Kaye SB, Schellens JH, de Bono JS. Inhibition of poly(ADP-ribose) polymerase in tumors from BRCA mutation carriers. N Engl J Med. 2009 Jul 9;361(2):123-34. doi: 10.1056/NEJMoa0900212. Epub 2009 Jun 24. PMID 19553641
- [Result] Tentori L, Lacal PM, Muzi A, Dorio AS, Leonetti C, Scarsella M, Ruffini F, Xu W, Min W, Stoppacciaro A, Colarossi C, Wang ZQ, Zhang J, Graziani G. Poly(ADP-ribose) polymerase (PARP) inhibition or PARP-1 gene deletion reduces angiogenesis. Eur J Cancer. 2007 Sep;43(14):2124-33. doi: 10.1016/j.ejca.2007.07.010. Epub 2007 Aug 21. PMID 17714938
- [Result] Bindra RS, Gibson SL, Meng A, Westermark U, Jasin M, Pierce AJ, Bristow RG, Classon MK, Glazer PM. Hypoxia-induced down-regulation of BRCA1 expression by E2Fs. Cancer Res. 2005 Dec 15;65(24):11597-604. doi: 10.1158/0008-5472.CAN-05-2119. PMID 16357170
- [Result] Bindra RS, Schaffer PJ, Meng A, Woo J, Maseide K, Roth ME, Lizardi P, Hedley DW, Bristow RG, Glazer PM. Down-regulation of Rad51 and decreased homologous recombination in hypoxic cancer cells. Mol Cell Biol. 2004 Oct;24(19):8504-18. doi: 10.1128/MCB.24.19.8504-8518.2004. PMID 15367671
- [Result] Lim JJ, Yang K, Taylor-Harding B, Wiedemeyer WR, Buckanovich RJ. VEGFR3 inhibition chemosensitizes ovarian cancer stemlike cells through down-regulation of BRCA1 and BRCA2. Neoplasia. 2014 Apr;16(4):343-53.e1-2. doi: 10.1016/j.neo.2014.04.003. PMID 24862760
- [Result] Liu JF, Tolaney SM, Birrer M, Fleming GF, Buss MK, Dahlberg SE, Lee H, Whalen C, Tyburski K, Winer E, Ivy P, Matulonis UA. A Phase 1 trial of the poly(ADP-ribose) polymerase inhibitor olaparib (AZD2281) in combination with the anti-angiogenic cediranib (AZD2171) in recurrent epithelial ovarian or triple-negative breast cancer. Eur J Cancer. 2013 Sep;49(14):2972-8. doi: 10.1016/j.ejca.2013.05.020. Epub 2013 Jun 27. PMID 23810467
- [Result] Liu JF, Barry WT, Birrer M, Lee JM, Buckanovich RJ, Fleming GF, Rimel B, Buss MK, Nattam S, Hurteau J, Luo W, Quy P, Whalen C, Obermayer L, Lee H, Winer EP, Kohn EC, Ivy SP, Matulonis UA. Combination cediranib and olaparib versus olaparib alone for women with recurrent platinum-sensitive ovarian cancer: a randomised phase 2 study. Lancet Oncol. 2014 Oct;15(11):1207-14. doi: 10.1016/S1470-2045(14)70391-2. Epub 2014 Sep 10. PMID 25218906
- [Result] Tan DS, Rothermundt C, Thomas K, Bancroft E, Eeles R, Shanley S, Ardern-Jones A, Norman A, Kaye SB, Gore ME. "BRCAness" syndrome in ovarian cancer: a case-control study describing the clinical features and outcome of patients with epithelial ovarian cancer associated with BRCA1 and BRCA2 mutations. J Clin Oncol. 2008 Dec 1;26(34):5530-6. doi: 10.1200/JCO.2008.16.1703. Epub 2008 Oct 27. PMID 18955455
- [Result] Birkbak NJ, Wang ZC, Kim JY, Eklund AC, Li Q, Tian R, Bowman-Colin C, Li Y, Greene-Colozzi A, Iglehart JD, Tung N, Ryan PD, Garber JE, Silver DP, Szallasi Z, Richardson AL. Telomeric allelic imbalance indicates defective DNA repair and sensitivity to DNA-damaging agents. Cancer Discov. 2012 Apr;2(4):366-375. doi: 10.1158/2159-8290.CD-11-0206. Epub 2012 Mar 22. PMID 22576213
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Lorusso D, Maltese G, Sabatucci I, Cresta S, Matteo C, Ceruti T, D'Incalci M, Zucchetti M, Raspagliesi F, Sonetto C, Sinno V, Ronzulli D, Giolitto S, de Braud F. Phase I Study of Rucaparib in Combination with Bevacizumab in Ovarian Cancer Patients: Maximum Tolerated Dose and Pharmacokinetic Profile. Target Oncol. 2021 Jan;16(1):59-68. doi: 10.1007/s11523-020-00780-4. Epub 2020 Dec 28. PMID 33369704